CLINICAL TRIAL: NCT00689949
Title: Determination of the Suitability of Urinary Total P-aminobenzoylglutamate (p-ABG)and Formiminoglutamate (FIGLU) as a Markers for Folate Status
Brief Title: Validation of Urinary Biomarkers of Folate Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: European Union (Other)
Responsible Party: Head of the Department for Nutrition and Metabolic Diseases, Haunersche Kinderklinik, Ludwig-Maximilians-University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 144-08
Record Dates: First submitted 2008-05-30; First posted 2008-06-04 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
Keywords: folic acid; folate; p-aminobenzoylglutamate; formiminoglutamate; homocysteine; experimental validation of a new biomarker
MeSH Terms: interventions — Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- folic acid (Other)
  Interventions: Dietary Supplement: folic acid

INTERVENTIONS:
Dietary Supplement: folic acid — 0.4 mg of folic acid per day

SUMMARY:
The major objective of the proposed study is to demonstrate the suitability of new markers for folate status in humans, which avoid blood sampling, as required for the established marker RBC folate concentration, but can be obtained from spot urine samples. For this reason urine and blood will be collected from volunteers, twice at baseline and in a subgroup after 6 and 12 weeks of intake of a folic acid supplement

Specific hypotheses to be tested:

Correlation study:

* The 24 h urinary excretion of total p-ABG, as extrapolated via urinary creatinine concentration from the total p-ABG concentration in a spot sample is significantly correlated to RBC and plasma folate levels in the studied subjects
* The 24 h urinary excretion of FIGLU, as extrapolated via urinary creatinine concentration form the FIGLU concentration in a spot sample is significantly correlated to RBC and plasma folate levels in the studied subjects

Intervention study:

Changes in folate status (RBC folate) after supplementary intake of folate result in increased urinary excretion of total p-ABG and FIGLU in subjects identified with a low folate status and in subjects identified with a high folate status among the study participants of the correlation study

ELIGIBILITY:
Inclusion Criteria:

* age: 18 - 45 years
* apparently healthy
* normal results on haematologic pattern and blood chemistry tests (according to university hospital reference values)
* plasma vitamin B12 > 160 pmol/l
* no diagnosis of intestinal, renal or thyroid disease (self reported)
* only male subjects will be enrolled but regular consumption of vitamin supplements (including folate) is not an exclusion criterium, as we aim to cover a wide range of folate concentrations.

Exclusion Criteria:

* recent (3 months) treatment with medication, assumed to interfere with folate status
* abuse of alcohol or drugs

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
correlation between red blood cell folic acid concentration and urinary excretion of total p-aminobenzoylglutamate | study day 1

SECONDARY OUTCOMES:
correlation between red blood cell folic acid concentration and urinary excretion of total p-aminobenzoylglutamate | study day 42
correlation between red blood cell folic acid concentration and urinary excretion of total p-aminobenzoylglutamate | study day 84

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Koletzko, Prof. Dr., Principal Investigator — Haunersche Kinderklinik, Ludwig-Maximilians-University
Locations (1):
- Haunersche Kinderklinik, München, Germany